CLINICAL TRIAL: NCT04238390
Title: A Multicentre, Parallel Group Open-label Randomised Controlled Non-Inferiority Phase 3 Trial, of Ceftolozane-tazobactam Versus Meropenem for Definitive Treatment of Bloodstream Infection Due to Extended-Spectrum Beta-Lactamase (ESBL) and AmpC-producing Enterobacterales
Brief Title: Ceftolozane-tazobactam Versus Meropenem for ESBL and AmpC-producing Enterobacterales Bloodstream Infection
Acronym: MERINO III
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The decision to withdraw the study was made due to delayed logistics of the supply chain of ceftolozane-tazobactam along with the immense complexities of conducting clinical research felt because of the COVID-19 pandemic.
Sponsor: The University of Queensland (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UQCCR-DP-AS-2019-001
Record Dates: First submitted 2019-12-16; First posted 2020-01-23 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2021-10

CONDITIONS: Bacteremia Caused by Gram-Negative Bacteria
MeSH Terms: interventions — ceftolozane, tazobactam drug combination; Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ceftolozane-tazobactam (Experimental): Participants will receive ceftolozane-tazobactam 3 grams (comprising ceftolozane 2 grams and tazobactam 1 gram) administered, every 8 hours, three times a day, intravenously over 60 mins
  Interventions: Drug: Ceftolozane-Tazobactam
- Meropenem (Active Comparator): Participants will receive meropenem 1 gram, every 8 hours, three times a day, intravenously over 30 mins.
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Ceftolozane-Tazobactam — Ceftolozane-tazobactam 3 grams (comprising ceftolozane 2 grams and tazobactam 1 gram) administered, every 8 hours, three times a day, intravenously over 60 mins. Dose adjusted for renal function.
  Arms: Ceftolozane-tazobactam
Drug: Meropenem — Meropenem 1 gram, every 8 hours, three times a day, intravenously over 30 mins. Dose adjusted for renal function.
  Arms: Meropenem

SUMMARY:
The purpose of this study is to determine whether ceftolozane-tazobactam is as effective as meropenem with respect to 30 day mortality in the treatment of bloodstream infection due to third-generation cephalosporin non-susceptible Enterobacterales or a known chromosomal AmpC-producing Enterobacterales (Enterobacter spp., Citrobacter freundii, Morganella morganii, Providencia spp. or Serratia marcescens).

DETAILED DESCRIPTION:
Enterobacterales are common causes of bacteraemia, and may produce extended-spectrum beta-lactamases (ESBLs) or AmpC beta-lactamases. ESBL or AmpC producers are typically resistant to third generation cephalosporins such as ceftriaxone, but susceptible to carbapenems. In no study has the outcome of treatment for serious infections for ESBL producers been significantly surpassed by carbapenems. Despite the potential advantages of carbapenems for treatment of ceftriaxone non-susceptible organisms, widespread use of carbapenems may cause selection pressure leading to carbapenem-resistant organisms. This is a significant issue since carbapenem-resistant organisms are treated with last-line antibiotics such as colistin.

Ceftolozane-tazobactam is a combination of a new beta-lactam antibiotic with an existing beta-lactamase inhibitor, tazobactam, and is active against ESBL and most AmpC producing organisms. In a large sample of ESBL- and AmpC-producing Enterobacterales isolates from urinary tract and intra-abdominal specimens, ceftolozane-tazobactam was susceptible in over 80%. It has been FDA approved for complicated urinary tract infections (cUTI) and complicated intra-abdominal infections (cIAI), and more recently for hospital-acquired and ventilator-associated pneumonia (HAP/VAP). In addition, a pooled analysis of phase 3 clinical trials has shown favourable clinical cure rates with ceftolozane-tazobactam for cUTI and cIAI caused by ESBL-producing Enterobacterales. Given the issues of carbapenem resistant organisms, there is a need for establishing the efficacy of an alternative to carbapenems for serious infections.

ELIGIBILITY:
Inclusion Criteria:

* Bloodstream infection defined as presence in at least one peripheral blood culture draw demonstrating Enterobacterales with proven non-susceptibility to third generation cephalosporins or cephalosporin susceptible species known to harbour chromosomal AmpC-beta-lactamases (Enterobacter spp., Klebsiella aerogenes, Citrobacter freundii, Morganella morganii, Providencia spp. or Serratia marcescens) during hospitalisation
* Patient is aged 18 years and over (21 and over in Singapore)
* The patient or approved proxy is able to provide informed consent
* ≤72 hours has elapsed since the first positive qualifying (index) blood culture collection
* Expected to receive IV therapy for ≥5 days

Exclusion Criteria:

* Known hypersensitivity to a cephalosporin or a carbapenem, or anaphylaxis to beta-lactam antibiotics
* Participant with significant polymicrobial bloodstream infection (i.e. not a contaminant)
* Treatment is not with the intent to cure the infection (i.e. palliative intent) or the expected survival is ≤4 days
* Participant is pregnant or breast-feeding (tested for in women of child-bearing age only)
* Use of concomitant antimicrobials with known activity against Gram-negative bacilli (except trimethoprim/sulfamethoxazole for Pneumocystis prophylaxis and when adding metronidazole for suspected IAI) in the first 5 days post-randomisation
* Participant with CrCl <15 mL/minute or on renal replacement therapy (in addition, participants will be withdrawn from the study if CrCl reaches this level)
* Previously randomised in the MERINO-3 trial or concurrently enrolled in another therapeutic antibiotic clinical trial
* Blood culture isolate with in-vitro resistance to either meropenem or ceftolozane-tazobactam (known either at time of enrolment or during the course of study treatment, in which case the participant will be withdrawn)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mortality rate at 30 days | 30 days post randomisation
  To compare the 30-day mortality from day of randomisation of each regimen

SECONDARY OUTCOMES:
Mortality rate at 14 days | 14 days post randomisation
  To compare the 14-day mortality from day of randomisation of each regimen
Clinical and microbiological success | 5 days post randomisation
  Defined as survival PLUS resolution of fever (temperature <38 degrees Celsius) PLUS improved SOFA score (as compared to baseline) PLUS sterilisation of blood cultures at Day 5
Functional bacteraemia score (FBS) | 0 and 30 days post randomisation
  To compare the functional bacteraemia score of patients treated with each regimen at baseline and Day 30 (scored 0-7, higher scores equal better outcomes)
Microbiological relapse | 30 days post randomisation
  To compare the rates of relapse of bloodstream infection (microbiological failure) with each regimen at Day 30
Rates of new bloodstream infection | 30 days post randomisation
  To compare the rates of new bloodstream infection (growth of a new organism from blood cultures - not a contaminant as determined by treating clinician) with each regimen
Length of in-patient hospital and ICU stay | 30 days post randomisation
  To compare lengths of in-patient hospital and ICU stay with each regimen (not including in-patient rehabilitation, long term acute care or hospital in the home)
Serious adverse events | Day 1 to last dose plus 24 hours of treatment:
  To compare the number of treatment emergent serious adverse events with each regimen
Clostridioides difficile infection | 30 days post randomisation
  To compare rates of Clostridioides difficile infection with each regimen
Colonisation and/or infection with multi-resistant bacterial organisms | 30 days post randomisation
  To compare rates of colonisation and/or infection with multi-resistant bacterial organisms (MROs) including those newly acquired
Desirability of Outcome Ranking (DOOR) with partial credit | 30 days post randomisation
  To compare the Desirability of Outcome Ranking (DOOR) with partial credit with each regimen (scored 0-100, higher scores equal better outcomes)

CONTACTS AND LOCATIONS:
Locations (29):
- Australia (13):
  - John Hunter Hospital, Newcastle, New South Wales
  - Royal Prince Alfred, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Woolongong Hospital, Wollongong, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Dandenong Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Sir Charles Gairdner, Perth, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia
- Italy (5):
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Dipartimento di Scienze Biomediche e Cliniche, Milan
  - Università di Pisa, Pisa
  - Policlinico Umberto, Roma
  - Sanremo Hospital, Sanremo
- Saudi Arabia (3):
  - King Fahad Specialist Hospital, Dammam
  - King Abdulaziz Medical City - Jeddah, Jeddah
  - King Abdulaziz Medical City, Riyadh
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- Spain (5):
  - Bellvitge University Hospital, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Sant Pau, Barcelona
  - Mutua Terrassa University Hospital, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stewart AG, Harris PNA, Chatfield MD, Littleford R, Paterson DL. Ceftolozane-tazobactam versus meropenem for definitive treatment of bloodstream infection due to extended-spectrum beta-lactamase (ESBL) and AmpC-producing Enterobacterales ("MERINO-3"): study protocol for a multicentre, open-label randomised non-inferiority trial. Trials. 2021 Apr 22;22(1):301. doi: 10.1186/s13063-021-05206-8. PMID 33888139